CLINICAL TRIAL: NCT06140095
Title: Studies to Gain Insight How the Drugs PCSK9-inhibitors and Statins Affect Cholesterol and Bile Acid Metabolism
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Stockholm (Other Government)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PSM1A
Record Dates: First submitted 2023-05-10; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-05

CONDITIONS: Acute Metabolic Effects of Evolocumab and Atorvastatin
MeSH Terms: interventions — evolocumab; Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Full group (Experimental): Evolocumab 140 mg subcutaneously. Två months later, repetitive doses of atorvastatin 40 mg once daily.
  After continued atorvastatin, evolocumab 140 mg is added subcutaneously.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — See arm description
  Other Names: Atorvastatin

SUMMARY:
Eight healthy male volunteers will be studied in consecutive sessions regarding the acute effect of evolocumab and atorvastatin on cholesterol and bile metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Male
* >18 years of age

Exclusion Criteria:

* Cardiovascular disease
* Cerebrovascular disease (e.g. stroke, prior aneurysm)
* Pulmonary disease (e.g. pulmonary hypertension, COPD)
* Metabolic disease (incl. but not limited to Cushing disease, Diabetes)
* Renal disease (by Chronic kidney disease criteria)
* Active inflammatory bowel syndrome
* Cancer
* Pregnancy
* Smoker
* Any chronic medication use
* Steroid treatment for the last six months or hormone replacement therapy
* Coagulopathy
* Musculoskeletal or neurologic disease
* Know allergy against any of the studied substances
* Inclusion in any other concurrent medical research study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cholesterol metabolism effect | 32 hours
  Effect of these treatments on markers for cholesterol metabolism, namely lathosterol and campesterol, measured as change from baseline concentration (mg/mmol) per unit time.
Bile acid metabolism effect | 32 hours
  Effect of these treatments on markers for bile acid metabolism, namely C4; measured as change from baseline concentration (mg/mmol) per unit time.
Bile acid metabolism effect | 32 hours
  Effect of these treatments on markers for cholesterol and bile acid metabolism, namely bile acids; measured as change from baseline concentration (mikromol/ml) per unit time.

IPD SHARING:
Plan to Share IPD: Undecided